CLINICAL TRIAL: NCT04276038
Title: Evaluation of the Efficacy of a Home-Use Photobiomodulation Device for the Treatment of Patients With Knee Osteoarthritis: A Prospective Double Blind, Randomized, Sham-Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, R&D deputy, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0438-19-TLV
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active LLLT (Active Comparator): Patients will self-treat at home (active or sham), twice a day (excluding Weekends) for 1 month. The duration of each session will be 15-20 minutes and will include treatment over painful point on the knee and over regional lymph nodes (popliteal, inguinal). The treatment dose should be initiated gradually for the first week until reaching the maximum dose of 6-8 minutes per treatment point. This is the recommended dose for near infrared lasers for the indication of knee pain by the World Association for Laser Therapy (WALT). In the first days an increase in pain may be felt before the reduction in pain. If the increase in pain continues for more than a week under graded dosimetry, the treatment must be stopped.
  Laser therapy will be administered to the patients in addition to standard of care therapy as customary in our institution.
  Interventions: Device: B-Cure laser pro
- Sham LLLT (Sham Comparator): Half of the LLT devices will be not activated at random before the application to the patients. Sham activated devices will give outward signs of normal function but will not generate a signal. The investigators will be unaware of the device's functionality. The patients will not be able to determine whether the device is working or not. At study completion, device serial numbers will be used to determine which patients received a working device.
  Interventions: Device: B-Cure laser pro

INTERVENTIONS:
Device: B-Cure laser pro — The B-Cure laser pro is a portal, non-invasive, low level laser therapy device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 1J/cm2. The device is used at home and is self-applied by the patient. The device is AMAR approved (approval # 14810408) for pain reduction and for ulcer treatment. The device is also approved for marketing in Canada and as a medical device in Europe (CE medical mark).

SUMMARY:
Osteoarthritis (OA) is a degenerative disease affecting joint cartilage and its surrounding tissue. It is the leading cause of disability in the elderly. The treatment of this disease remains limited to symptomatic relief and, ultimately, joint replacement. Despite the progress made in understanding the pathophysiology of OA, effective disease-modifying drugs are still lacking.

Low-level laser therapy (LLLT), also known as Photobiomodulation therapy, is a non-ionizing optical radiation in the visible or near infrared range of the spectrum. LLLI has been used widely for alleviation of pain, reduction of inflammation, and acceleration of wound healing. Specifically, it has been shown to reduce pain in chronic inflammatory related knee pathologies in pre-clinical and clinical studies. However, the recommended treatment protocol requires frequent treatments that translates to frequent visits at the clinic. Such a treatment regimen is difficult for Knee OA (KOA) patients and demanding of the clinical staff. Since the treatment itself can be self-applied easily, a home-use device would enable frequent treatments thereby improving patient adherence to the treatment.

In a pilot study, Kruglova et al [4] reported that 2 weeks of daily treatments with the home use B-Cure laser significantly reduced pain and increased flexibility in 20 elite athletes with KOA.

The purpose of the current study is to determine if B-Cure laser treatments, applied at home, by the patient or personal caregiver in a real-life situation, can reduce pain and improve functionality in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of knee osteoarthritis:( American College of Rheumatology (ACR) criteria (see below) - possibilities:ACR1: Fulfilled at least one of the classification criteria of the American College of Rheumatology ACR2: KOA verified with the American College of Rheumatology criteria using a history and physical examination, i.e. knee pain and at least three of the following: 50-85 years old, ≤ 30 minutes of morning stiffness, crepitus on active range of motion, bony tenderness, bony enlargement, and no palpable warmth of synovia Radiographic evidence of knee osteoarthritis between 2-3 in Kellgren and Lawrence classification
* KOA grade 2-3
* Knee pain on movement 40 to 90 mm Visual Analog Scale
* Knee pain for the last ≥ 3 months
* Functional reduction in the last three months
* Agrees not to use NSAIDs throughout the experiment
* Agrees not to use any other treatment (except rescue drugs) for KOA during participation in this study.

Exclusion Criteria:

* Other causes of knee-related pain (e.g. hip OA, arterial insufficiency, etc) have been ruled out by physical examinations
* Knee surgery for KOA
* Intra-articular steroid injection and/or oral steroid treatment within the last six months
* Rheumatoid arthritis;
* Symptomatic OA in other joints (i.e. hip, hand)
* Use of analgesics on the day of evaluation
* Use of NSAIDs 2 weeks before the beginning of the treatment
* Active malignancy
* Uncontrolled diabetes mellitus
* Neurological conditions: sciatica, neuropathy, multiple sclerosis
* Other chronic pain conditions: Fibromyalgia, back pain, hip pain
* Enrolled in any other clinical trial within the last 6 weeks or enrollment in another clinical trial during participation in this trial.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of B-cure laser for pain reduction in patients with knee osteoarthritis | time point - 1 month
  Change from baseline in pain score by visual analog scale (VAS), 0-10, 0 - no pain; 10- worst pain

SECONDARY OUTCOMES:
Range of Movement | time point - 1 month
  Change from baseline

IPD SHARING:
Plan to Share IPD: No